CLINICAL TRIAL: NCT00435123
Title: A Randomized, Placebo Controlled, Double Blind Study of the Use of a Nutritional Supplement, ProStat-64, in Chronic Hemodialysis Patients With Poor Nutritional Status.
Brief Title: ProStat Supplementation in Dialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Increased use of commercial product; less eligible patients & poor enrollment.
Sponsor: Fresenius Medical Care North America (Industry)
Collaborators: Medical Nutrition USA, Inc. (Industry)
Responsible Party: Mark Kaplan, M.D., Vice-President Research, Fresenius Medical Care North America
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006002; 061201 Vanderbilt IRB; NCT00458939 (obsolete NCT alias)
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Malnutrition; ESRD
Keywords: Malnutrition; ESRD; Hemodialysis
MeSH Terms: conditions — Malnutrition; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Patients are randomly assigned to receive either Active Comparator (ProStat 64) or placebo for the first 3 months. At the end of this, all patients receive open label ProStat64.
  Interventions: Dietary Supplement: Nutritional Supplement ProStat 64 twice a day
- B (Placebo Comparator): Patients are randomly assigned to Placebo Comparator or Active Comparator (ProStat 64). At the end of 3 months, all patients receive active ProStat 64
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement ProStat 64 twice a day
  Arms: A
Dietary Supplement: Placebo supplement — Patients randomly assigned to Placebo for the first 3 months will receive open label Prostat for the last 3 months
  Arms: B

SUMMARY:
This is a long-term, randomized, placebo-controlled, double blind clinical study of a nutritional supplement, ProStat 64, in chronic hemodialysis patients with poor nutrition. Subjects receive either ProStat 64 or Placebo for three months. At the end of this period, all subjects will receive ProStat-64 for a further 3 months at which time the study is ended. Parameters of nutritional status (lean body mass and serum protein) will be collected at baseline, 3 months and 6 months.

DETAILED DESCRIPTION:
Fifty patients identified as having poor nutrition by the following criteria:

1. Average of Serum Albumin for the consecutive two months prior to inclusion </= 3.7 g/dl and the serum albumin for the previous month is < 3.7 mg/dl.
2. one of the four following criteria:

   1. Protein catabolic rate less than 1.0 g/kg/d on at least 2 occasions over the past 6 months
   2. Progressive unintentional weight loss more than 2.5% of the initial or ideal body weight and/or patients who are less than 90% of Standard Body Weight
   3. Subjective Global Assessment Score consistent with Moderate to Severe Malnutrition within the last month
   4. Biochemical parameters of malnutrition defined by 1 of 2 of the following measurements (if available) over the consecutive two months prior to inclusion:

      1. Serum transferrin concentration less than 225 mg/dl
      2. Serum prealbumin concentration less than 32 mg/dl

will be randomized to receive either ProStat 64 or placebo for 3 months. At Baseline a Dexa for lean body mass and labs for BUN, creatinine, glucose, serum albumin, prealbumin and C-reactive protein will be drawn. Cholesterol and transferrin will be recorded from the regular monthly labs if available. In addition, a protein catabolic rate will be calculated and a SGA will be completed.

Patients will take the supplement/placebo twice a day. Measurements will be repeated at month 3. At the end of these measurements, all patients will be switched to open label ProStat64 for an additional 3 months. At month 6 all study procedures/labs are repeated and the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis
* Optimally dialyzed with a biocompatible membrane (URR > 70% and/or delivered Kt/V >1.2)
* Patient or next of kin able to sign consent form
* Average of Serum Albumin for the consecutive two months prior to inclusion </= 3.7 g/dl and the serum albumin for the previous month is < 3.7 mg/dl.
* Sub-optimal nutritional status identified by one of the four following criteria:

  1. Protein catabolic rate less than 1.0 g/kg/d on at least 2 occasions over the past 6 months
  2. Progressive unintentional weight loss more than 2.5% of the initial or ideal body weight and/or patients who are less than 90% of Standard Body Weight
  3. Subjective Global Assessment Score consistent with Moderate to Severe Malnutrition within the last month
  4. Biochemical parameters of malnutrition defined by 1 of 2 of the following measurements (if available) over the consecutive two months prior to inclusion:

     1. Serum transferrin concentration less than 225 mg/dl
     2. Serum prealbumin concentration less than 32 mg/dl
* Patient is able to transfer with minimal or no assistance.
* Not taking a caloric nutritional supplement for the last 30 days (e.g. Nepro, ProStat, Boost,etc).

Exclusion Criteria:

* Active auto-immune, inflammatory or infectious disease
* Documented malignancy within the last 12 months
* Patients on unusual dietary restrictions
* Life-expectancy less than 6 months
* Inability to tolerate nutritional supplements
* Patient does not exceed the DEXA machine weight limit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Increase in visceral protein stores as measured by serum albumin | 3 months minimum; 6 months max

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kaplan, M.D., Principal Investigator — Fresenius Medical Care North America; Alp Ikizler, M.D., Principal Investigator — Vanderbilt University
Locations (6):
- United States (6):
  - Kansas Nephrology Physicians, PA, Wichita, Kansas
  - Western New England Renal Transplant Associates, Springfield, Massachusetts
  - Nephrology Associates, Columbus, Mississippi
  - Midwest Nephrology Associates, City of Saint Peters, Missouri
  - Metro Hypertension & Kidney Center, LLC., St Louis, Missouri
  - Lankenau Center for Medical Research, Wynnewood, Pennsylvania

REFERENCES:
- [Background] Ikizler TA, Wingard RL, Harvell J, Shyr Y, Hakim RM. Association of morbidity with markers of nutrition and inflammation in chronic hemodialysis patients: a prospective study. Kidney Int. 1999 May;55(5):1945-51. doi: 10.1046/j.1523-1755.1999.00410.x. PMID 10231458
- [Background] Ikizler TA, Hakim RM. Nutrition in end-stage renal disease. Kidney Int. 1996 Aug;50(2):343-57. doi: 10.1038/ki.1996.323. PMID 8840260
- [Background] Caglar K, Fedje L, Dimmitt R, Hakim RM, Shyr Y, Ikizler TA. Therapeutic effects of oral nutritional supplementation during hemodialysis. Kidney Int. 2002 Sep;62(3):1054-9. doi: 10.1046/j.1523-1755.2002.00530.x. PMID 12164890
- [Background] Pupim LB, Flakoll PJ, Brouillette JR, Levenhagen DK, Hakim RM, Ikizler TA. Intradialytic parenteral nutrition improves protein and energy homeostasis in chronic hemodialysis patients. J Clin Invest. 2002 Aug;110(4):483-92. doi: 10.1172/JCI15449. PMID 12189242